CLINICAL TRIAL: NCT05882136
Title: Assessment of the Structure and Function of Heart and Selected Cardiovascular Risk Factors in Patients With Acute Intermittent Porphyria
Brief Title: Acute Intermittent Porphyria Related Abnormalities in Cardiovascular System
Acronym: AIPRACUS
Status: Completed | Type: Observational
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Collaborators: Institute of Hematology and Transfusion Medicine, Warsaw (Other)
Responsible Party: Principal Investigator, Krzysztof Jaworski, Principal Investigator, National Institute of Cardiology, Warsaw, Poland
Other Study IDs: 2.39/VII/18
Record Dates: First submitted 2023-05-03; First posted 2023-05-31 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Porphyrias, Hepatic
Keywords: acute intermittent porphyria; myocardial injury; heart failure; hypertension; cardiac arrhythmia; cardiovascular risk factors; lipid profile; quality of life
MeSH Terms: conditions — Porphyrias, Hepatic; Porphyria, Acute Intermittent; Heart Failure; Hypertension; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with acute intermittent porphyria (AIP): Patients aged 18-65 (men and women) with acute intermittent porphyria and at least one episode of exacerbation of this disease requiring admission to the hospital
- Control group: People recruited from the general population and matched by age, sex and body mass index.

SUMMARY:
This study aims to assess the changes in the cardiovascular system in patients with acute intermittent porphyria (AIP).

DETAILED DESCRIPTION:
Porphyrias are heterogeneous group of the disorders of heme biosynthesis. Acute intermittent porphyria (AIP) is the most common acute hepatic porphyria, caused by the mutations in the gene encoding hydroxymethylbilane synthase. Clinical symptoms i.e. abdominal pain, nausea, vomiting, paresis or paralysis, coma and/or mental abnormalities may be induced by many porphyrinogenic factors, such as drugs, alcohol, starvation or stress. The symptoms are often accompanied by tachycardia and elevated blood pressure. Due to the non-specific clinical picture, AIP is often diagnosed too late and causes a threat to the patients' lives.

There is a scarcity of data regarding the changes in cardiovascular system in patients with AIP. The aim of this study is to assess the structure and function of heart in patients with this disease. The prevalence of hypertension, cardiac arrhythmias and selected cardiovascular risk factors in patients with AIP will also be evaluated.

This is a case-control study with prospective observation of the subgroup of patients examined during the exacerbations of AIP.

Specific goals:

* assessment of the cardiac morphology and function,
* assessment of the concentrations of markers of myocardial injury (troponin T) and heart failure (NT-proBNP),
* assessment of the prevalence of cardiac arrhythmias and electrocardiographic abnormalities,
* assessment of the blood pressure profiles,
* assessment of selected cardiovascular risk factors,
* assessment of quality of life,
* assessment of clinical and biochemical factors associated with the pathological findings in patients with AIP.

ELIGIBILITY:
Inclusion Criteria:

* acute intermittent porphyria (AIP),
* age 18-65 years,
* at least one hospitalization due to exacerbation of AIP.

Exclusion Criteria:

* previous myocardial infarction,
* heart failure of established (other than porphyria) etiology,
* severe heart valve disease,
* congenital heart defects,
* history of myocarditis,
* pacemaker,
* hyperthyroidism / hypothyroidism (except for adequate thyroid hormone replacement therapy),
* chronic advanced lung diseases,
* lack of consent to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients with acute intermittent porphyria (AIP) meeting the eligibility criteria and people from the general population, matched by age, sex and body mass index.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with heart failure and left ventricular dysfunction. | day 1 and up to 2 years in case of the exacerbation of AIP
  Heart failure and left ventricular dysfunction assessed by symptoms and echocardiography.
Number of participants with hypertension. | day 1 and up to 2 years in case of the exacerbation of AIP
  Arterial hypertension diagnosed by ambulatory 24-hour blood pressure monitoring.
Rate of cardiac arrhythmias. | day 1 and up to 2 years in case of the exacerbation of AIP
  Cardiac arrhythmias observed in 24-hour ECG monitoring.

SECONDARY OUTCOMES:
Number of participants with increased concentrations of markers of heart failure. | day 1 and up to 2 years in case of the exacerbation of AIP
  Concentration of N-terminal pro-B-type natriuretic peptide (NT-proBNP) > 125 pg/mL in serum.
Number of participants with increased concentrations of markers of myocardial injury. | day 1 and up to 2 years in case of the exacerbation of AIP
  Concentration of high sensitivity troponin T > 14 ng/L in serum.
Number of participants with chronic kidney disease. | day 1 and up to 2 years in case of the exacerbation of AIP
  Renal function defined by estimated glomerular filtration rate based on the concentrations of creatinine in serum.
Number of participants with dyslipidemia. | day 1
  Dyslipidemia defined as the concentrations of total cholesterol > 190 mg/dL, low density lipoprotein (LDL) cholesterol > 115 mg/dL, high density lipoprotein (HDL) cholesterol < 48 mg/dL (female), < 40 mg/dL (male), triglycerides > 150 mg/dL.
Number of participants with diabetes. | day 1
  Diabetes in anamnesis or the concentration of glycated hemoglobin > 6.5%.
Level of quality of life. | day 1
  Physical and mental components defined by the Short Form 36 survey (SF36). Answers are weighted and transformed into scores in a scale ranging from 0 (the lowest possible level of functioning) to 100 (no restrictions).

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Jaworski, MD, Principal Investigator — National Institute of Cardiology, Warsaw, Poland
Locations (2):
- Poland (2):
  - Institute of Hematology and Transfusion Medicine, Warsaw
  - National Institute of Cardiology, Warsaw

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jaworski K, Wasilewski R, Windyga J, Januszewicz A, Szwed H, Dabrowski R. Cardiovascular abnormalities in patients with acute intermittent porphyria: the AIPRACUS study. Pol Arch Intern Med. 2024 Aug 8;134(7-8):16820. doi: 10.20452/pamw.16820. Epub 2024 Aug 8. No abstract available. PMID 39115302